CLINICAL TRIAL: NCT06284083
Title: COMPARİSON OF AGMATİNE, TELOMERASE, AND SOME TRACE ELEMENT LEVELS İN PATİENTS WİTH DİFFERENT SEVERİTY OF OBSTRUCTİVE SLEEP APNEA SYNDROME. Start Date: 18.12.2018
Brief Title: Measuring Various Variables in Obstructive Sleep Apnea
Acronym: OUAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Dilara Ulger Ozbek, Ph.D,main investigator, Cumhuriyet University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Cumhuriyet University Hospital
Record Dates: First submitted 2022-08-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: sleep apnea; agmatine; telomerase; trace elements
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: The study group consisted of 90 newly diagnosed OSAS patients who were admitted to the Clinic for Chest Diseases of the Research and Practice Hospital of Sivas Cumhuriyet University Faculty of Medicine. For the definitive diagnosis of OSAS, the patients were hospitalized overnight in the Sleep Center and polysomnography test was performed. OSAS patients, who were randomly selected without discrimination in terms of age and gender, were connected to the PSG device for one night and various measurements were taken and the values were recorded. The apnea/hypopnea index (AHI) was defined as the sum of the apnea and hypopnea number per hour of sleep. Volunteer patients were grouped into three based on apnea-hypopnea index (AHI) scores: mild OSAS (n=30; 5 ≤ AHI ≤ 13.70), moderate (n=30; 15.80 ≤ AHI ≤ 26.60) and severe (n=30; 34.10 ≤ AHI ≤ 86.30). The mean SpO2 percentages of the PSG device were measured from the fingertip with a system-defined pulse oximeter.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polysomnographic (PSG) diagnosis and scoring.Oxygen saturation mesurment (SpO2) (No Intervention): The participants were put to sleep with polysomnography (PSG) in the sleep laboratory for 1 night and were divided into 3 groups according to their disease severity. (mild, moderate, severe).The apnea/hypopnea index (AHI) was defined as the sum of the apnea and hypopnea number per hour of sleep. The mean SpO2 percentages of the PSG device were measured from the fingertip with a system-defined pulse oximeter.
- Agmatine, Telomerase and Trace element levels measurment (Experimental): With the permission of the participants, 7 ml of venous, fasting blood was taken after the night's sleep.In the blood serum of the participants, agmatine, telomerase, and trace element levels were measured with a commercial ELISA kit.
  Interventions: Diagnostic Test: taking a blood sample

INTERVENTIONS:
Diagnostic Test: taking a blood sample — Blood samples collected from patienst, only 7 mL
  Arms: Agmatine, Telomerase and Trace element levels measurment

SUMMARY:
This study included 90 volunteer Obstructive Sleep Apnea Syndrome patients. Only 7 mL blood samples collected from patients. Some biochemicals parameters analyzed in blood serum/plasma.

DETAILED DESCRIPTION:
This study included 90 volunteer patients diagnosed with OSAS, and they were divided into three groups according to the apnea-hypopnea index (AHI) score: mild OSAS (n=30;5≤ AHI ≤13.70), moderate (n=30;15.80≤AHI≤26.60) and severe (n=30;34.10≤AHI≤86.30). Demographic data, as well as biochemical parameters, nocturnal oxygen saturation percentage (SpO2), and body mass index (BMI) were measured. Plasma agmatine levels were measured by ultra-high-pressure liquid chromatography (UHPLC), plasma trace elements (Cu, Co, Mg, Mo, Zn, Se) levels were determind by inductively coupled plasma mass spectrometer (ICP-MS) and serum telomerase levels were measured by enzyme-linked immunosorbent assay (ELISA) method. Analyzes were carried out at the Cumhuriyet University advanced technology research and application center.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obstructive sleep apnea disease
* Apnea-hypopnea index (AHI) score between 5-87

Exclusion Criteria:

* asthma
* chronic obstructive pulmonary disease
* pneumonia
* psychiatric
* diabetes
* heart failure
* who work at night work

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Agmatine, telomerase and trace element levels in blood serum vary depending on disease severity. | not measured in time frame. general (one day)
  Agmatine Telomerase and trace element levels will be measured in blood serum. The most common side effect when blood is taken from the patient is slight bruising and swelling in the arm due to needle sticking. There will be no other serious side effects.

SECONDARY OUTCOMES:
Polysomnographic measurement | one day
  Patients will be put to sleep for 1 night with polysomnography, and the severity of the disease will be determined by calculating the number of times breathing stops during sleep with the Apnea-hypoapnea index. There will be no side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Sevtap BAKIR, Professor, Study Chair — Cumhuriyet University; Ömer Tamer DOĞAN, Professor, Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Centre, Turkey (Türkiye)